CLINICAL TRIAL: NCT04401345
Title: Effect of Glycopyrrolate on Vasopressors Requirement for Non-elective Caesarean Section Under Spinal Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rajesh Deshar (Other)
Responsible Party: Sponsor-Investigator, Rajesh Deshar, Principal Investigator, B.P. Koirala Institute of Health Sciences
Organization: B.P. Koirala Institute of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRC/1603/019
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Glycopyrrolate; Post-spinal Hypotension; Effect of Drug; Hemodynamic Instability
Keywords: caesarean section; hypotension; spinal anaesthesia; glycopyrrolate; post-spinal anaesthesia; vasopressors; non-elective caesarean section
MeSH Terms: conditions — Hypotension | interventions — Glycopyrrolate; Saline Solution

STUDY DESIGN:
Intervention Model Description: Experimental Group (GP): In the experimental group patients will receive 0.2 mg (1 ml) glycopyrrolate before phenylephrine infusion is initiated.
  Placebo Group (NS): In the placebo group patients will receive 1 ml normal saline (0.9%) before phenylephrine infusion is initiated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Glycopyrrolate and normal saline will be administered as 1 ml clear fluid, and therefore, both patient and investigator will be blinded to the randomization and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (GP) (Experimental): Patients will receive 0.2 mg (1 ml) glycopyrrolate before phenylephrine infusion is initiated at 25mcg/min.
  Interventions: Drug: Glycopyrrolate 0.2 MG/ML
- Placebo Group(NS) (Placebo Comparator): patients will receive 1 ml normal saline (0.9%) before phenylephrine infusion is initiated at 25 mcg/min
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Glycopyrrolate 0.2 MG/ML — In this group, the patients will receive glycopyrrolate 0.2 mg in 1 ml
  Other Names: Glycopyrronium bromide
  Arms: Experimental Group (GP)
Drug: Normal saline — In this group, the patients will receive 1 ml of 0.9% normal saline
  Other Names: 0.9% NS
  Arms: Placebo Group(NS)

SUMMARY:
This is prospective randomised double blind study conducted in parturients planned for non-elective caesarean section under spinal anaesthesia. Glycopyrrolate group will receive 0.2 mg of Glycopyrrolate before start of phenylephrine infusion. Control group will receive 0.2 ml of Normal Saline before start of phenylephrine infusion. Total amount of vasopressors required i.e. ephedrine or phenylephrine will recorded in the form of phenylephrine equivalent during intraoperative period.

DETAILED DESCRIPTION:
Intravenous glycopyrrolate has been investigated for its effect on haemodynamic changes after spinal anesthesia for caesarean delivery. Results from previous studies are conflicting as glycopyrrolate has shown to reduce, increase or had no effect on incidence of maternal hypotension and/or vasopressor requirement after spinal anaesthesia. A recent meta-analysis found that prophylactic glycopyrrolate does not prevent the incidence of spinal-induced hypotension; however, it reduces the total vasopressor requirement during elective caesarean delivery under spinal anaesthesia. Therefore, the aim of this study is to find out whether the use of glycopyrrolate decreases the amount of vasopressors required to manage hypotension induced by spinal anaesthesia in non-elective CS.

Methodology:

After approval from Institutional Review committee of B.P. Koirala Institute of Health Sciences, the trial will be registered at clinical trial.gov. Parturient planned for non-elective caesarian of ASA PS grade II fulfilling the inclusion criteria will be informed about the study and written consent will be obtained either in labour room or in obstetric emergency ward. The eligible patients will be randomly assigned to Glycopyrrolate (GP group) or normal saline (NS group). The study will be conducted in accordance with the ethical principles of the 1964 Declaration of Helsinki. Before patient is shifted to the operating room (OR), ranitidine 50 mg and metoclopramide 10 mg will be administered intravenously via 18 G cannula. In the operating table, patients will be laid supine with a wedge placed in the right hip. Standard anaesthesia monitoring including 3-lead electrocardiography, heart rate (HR), noninvasive blood pressure (NIBP) and pulse oximetry (Sp02) will be done. A mean value of three measurements of systolic blood pressure (SBP) and HR will be recorded as baseline parameters. Patency of the vein will be maintained with the infusion of Ringer's lactate solution at a minimal rate.

Before the patient is placed in sitting position for SA,she will receive the study drug according to the randomization. After free flow of CSF is observed, 0.5 % hyperbaric bupivacaine (2.2 ml) with 10 µg fentanyl will be injected intrathecally over 30 s using a 25-gauge Quinke needle at the L3-4 or L4-L5 interspace. Patients will then be immediately placed in supine while maintaining 15 degree left lateral tilt. Co-loading of 1000 ml ringers lactate solution will be initiated at the start of spinal anaesthesia using a pressure bag and it will be completed within 10 min. Immediately after the spinal injection, phenylephrine infusion will be initiated at a rate of 25 µg/min and it will be titrated to maintain maternal SBP within 20 % of baseline.

The sensory level of anaesthesia will be checked using loss of cold sensation. Surgery will be allowed once the bilateral sensory block height at T6 is achieved. Oxygen at 40% will be administered via nasal cannula at 2-4 L/min until delivery.

Hemodynamic parameters will be recorded at following time intervals: baseline, after the study drug in given IV, immediately after spinal anaesthesia, every minute for first 10 min, and then at 2.5 min until end of surgery. Post-spinal hypotension will be defined as SBP < 80% of baseline reading or SBP < 100 mmHg before delivery of baby. Post-delivery hypotension is defined as SBP < 80% of baseline reading or SBP < 100 mmHg after delivery of the baby. It will be treated with phenylephrine 100 µg bolus and rapid infusion of Ringer's lactate 200 ml. Infusion of phenylephrine will be stopped if bradycardia (HR< 55/min) occurs without hypotension. If bradycardia (HR< 55/min) is associated with hypotension, IV ephedrine 6 mg will be administered. If these measures fail and bradycardia is still persistent then an IV atropine 0.5 mg will be given. If reactive hypertension (defined as SBP > 120% of baseline reading) occurs, the infusion of phenylephrine will be stopped and restarted only when the SBP reaches the target range (SBP is within 120% of baseline SBP). The amount of ephedrine used will be converted to phenylephrine equivalent based on potency of phenylephrine to ephedrine as 81:1 ratio.(31)

After delivery of the baby, 2 U of oxytocin will be administered IV over 5-10 sec followed by an infusion of 10 U/hr (oxytocin 20 U in 500 ml of Hartmann's solution). Phenylephrine infusion will be gradually tapered after delivery of the baby keeping the SBP within the target level. The total amount of intraoperative IV fluids administered and estimated blood loss will be measured. Intraoperative use of other uterotonic agent or blood transfusion will be recorded. The attending pediatrician will assess neonatal Apgar scores at 1 and 5 minutes after delivery.

Patients will be asked to report the occurrence of intraoperative nausea and rate its severity using an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea). Intraoperative nausea or vomiting (IONV) will be treated with ondansetron 4 mg IV. After 5 min, if nausea and vomiting is still persisted, IV dexamethasone 4 mg will be administered. IONV incidence and its time of occurrence from intrathecal injection (whether associated with hypotension) and antiemetic needed will be recorded. Incidence of intraoperative pruritus, shivering, dizziness and dry mouth will also be recorded. Grading of intraoperative shivering is as follows: 0 no shivering, 1 one or more of the following: piloerection, peripheral vasoconstriction, peripheral cyanosis without other cause, but without visible muscular activity; 2 visible muscular activity confined to one muscle group; 3 visible muscular activity in more than one muscle group; and 4 gross muscular activity involving the whole body. If the shivering score is ≥3, IV meperidine 20 mg will be given.

The primary outcome will be the total amount of phenylephrine used to maintain blood pressure intraoperatively. The secondary outcome measures will include incidence of maternal hypotension, reactive hypertension, bradycardia, other side-effects (IONV, shivering, pruritus, dry mouth,dizziness), changes in maternal SBP and heart rate and neonatal outcome (Apgar scores at 1 min and 5 min, requirement of neonatal resuscitation, need for neonatal ICU admission and neonatal death within 30 days).

Data collection:

Baseline data (gestational age, uterine incision to delivery time, hemodynamic parameters) and outcome parameters will be collected in the paper case record form and entered in windows Microsoft excel spreadsheet for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years
* All parturients at term (gestational weeks ≥ 37)
* ASA (American society of Anaesthesiologist) PS (Physical status) grade II

Exclusion Criteria:

* Age >40 year
* ASA PS Grade >2
* Maternal bradycardia (baseline HR< 60/min) or tachycardia (baseline HR> 100/min)
* Pregnancy induced hypertension
* Gestational hypertension
* Known fetal abnormalities
* Intrauterine growth retardation (IUGR)
* Intrauterine fetal death (IUFD)
* Contraindications to spinal anaesthesia
* Contraindications to glycopyrrolate
* Multiple pregnancy
* BMI: > 30 kg/m2
* Height: <150cm

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Total vasopressors requirement intraoperatively | immediately after spinal anaesthesia till the end of the surgery
  Total vasopressors required to prevent hypotension during the period of surgery

SECONDARY OUTCOMES:
The incidence of hypotension | after spinal anaesthesia till the end of the surgery
  Hypotension is defined as systolic blood pressure < 80% of baseline reading or systolic blood pressure < 100 mmHg
The incidence of reactive hypertension | after spinal anaesthesia till the end of the surgery
  defined as systolic blood pressure > 120% of baseline reading
The incidence of maternal bradycardia | after spinal anaesthesia till the end of the surgery
  heart rate < 55/min
The incidence of maternal tachycardia | after spinal anaesthesia till the end of the surgery
  Heart rate > 100/min
The incidence of nausea | after spinal anaesthesia till the end of the surgery
  Patients will be asked to report the occurrence of intraoperative nausea and rate its severity using an 11-point verbal rating scale (0=no nausea, 10=worst possible nausea).
The incidence of vomiting | after spinal anaesthesia till the end of the surgery
  incidence of vomiting
The incidence of shivering | after spinal anaesthesia till the end of the surgery
  Shivering will be graded as: 0 no shivering, 1 one or more of the following: piloerection, peripheral vasoconstriction, peripheral cyanosis without other cause, but without visible muscular activity; 2 visible muscular activity confined to one muscle group; 3 visible muscular activity in more than one muscle group; and 4 gross muscular activity involving the whole body
The incidence of dry mouth, intraoperative pruritus and dizziness | after spinal anaesthesia till the end of the surgery
  incidence of dry mouth, intraoperative pruritus and dizziness
Maternal heart rate and | after spinal anaesthesia till the end of the surgery
  to record the heart rate of the patient during surgery
Maternal systolic blood pressure | after spinal anaesthesia till the end of the surgery
  to record systolic blood pressure of the patient during surgery

OTHER OUTCOMES:
The APGAR outcome of baby | at 1 and 5 min after delivery
  APGAR score comprises of 5 criteria : a) Appearance b) Pulse Rate c) Reflex d)Muscle tone e) Respiratory Effort with each criteria of score 0,1 or 2; making total score of 10. Score 7-10 is reassuring, 4-6 moderately normal, 0-3 is low and cause for immediate resuscitative efforts
Need for neonatal resuscitation | immediately after delivery
  resuscitation needed for baby
Admission to neonatal ICU (NICU) | after delivery
  the need for ICU admission
Neonatal death | within 30 days of delivery
  if there is neonatal death or not

CONTACTS AND LOCATIONS:
Locations (1):
- B.P.Koirala Institute of Health Sciences, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yentis SM, Jenkins CS, Lucas DN, Barnes PK. The effect of prophylactic glycopyrrolate on maternal haemodynamics following spinal anaesthesia for elective caesarean section. Int J Obstet Anesth. 2000 Jul;9(3):156-9. doi: 10.1054/ijoa.1999.0376. PMID 15321086
- [Background] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Result] Somboonviboon W, Kyokong O, Charuluxananan S, Narasethakamol A. Incidence and risk factors of hypotension and bradycardia after spinal anesthesia for cesarean section. J Med Assoc Thai. 2008 Feb;91(2):181-7. PMID 18389982
- [Result] Dyer RA, Biccard BM. Ephedrine for spinal hypotension during elective caesarean section: the final nail in the coffin? Acta Anaesthesiol Scand. 2012 Aug;56(7):807-9. doi: 10.1111/j.1399-6576.2012.02719.x. No abstract available. PMID 22780437
- [Result] Kinsella SM, Tuckey JP. Perioperative bradycardia and asystole: relationship to vasovagal syncope and the Bezold-Jarisch reflex. Br J Anaesth. 2001 Jun;86(6):859-68. doi: 10.1093/bja/86.6.859. PMID 11573596
- [Result] Dobson PM, Caldicott LD, Gerrish SP, Cole JR, Channer KS. Changes in haemodynamic variables during transurethral resection of the prostate: comparison of general and spinal anaesthesia. Br J Anaesth. 1994 Mar;72(3):267-71. doi: 10.1093/bja/72.3.267. PMID 8130043
- [Result] Ali S, Athar M, Ahmed SM. Basics of CPB. Indian J Anaesth. 2019;49:257-62.
- [Result] Lee AJ, Landau R. Aortocaval Compression Syndrome: Time to Revisit Certain Dogmas. Anesth Analg. 2017 Dec;125(6):1975-1985. doi: 10.1213/ANE.0000000000002313. PMID 28759487
- [Result] Dick WF. Anaesthesia for caesarean section (epidural and general): effects on the neonate. Eur J Obstet Gynecol Reprod Biol. 1995 May;59 Suppl:S61-7. doi: 10.1016/0028-2243(95)02075-4. PMID 7556827
- [Result] Kuhn JC, Hauge TH, Rosseland LA, Dahl V, Langesaeter E. Hemodynamics of Phenylephrine Infusion Versus Lower Extremity Compression During Spinal Anesthesia for Cesarean Delivery: A Randomized, Double-Blind, Placebo-Controlled Study. Anesth Analg. 2016 Apr;122(4):1120-9. doi: 10.1213/ANE.0000000000001174. PMID 26991619
- [Result] Cyna AM, Andrew M, Emmett RS, Middleton P, Simmons SW. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002251. doi: 10.1002/14651858.CD002251.pub2. PMID 17054153
- [Result] Lee AJ, Landau R, Mattingly JL, Meenan MM, Corradini B, Wang S, Goodman SR, Smiley RM. Left Lateral Table Tilt for Elective Cesarean Delivery under Spinal Anesthesia Has No Effect on Neonatal Acid-Base Status: A Randomized Controlled Trial. Anesthesiology. 2017 Aug;127(2):241-249. doi: 10.1097/ALN.0000000000001737. PMID 28598894
- [Result] Ripolles Melchor J, Espinosa A, Martinez Hurtado E, Casans Frances R, Navarro Perez R, Abad Gurumeta A, Calvo Vecino JM. Colloids versus crystalloids in the prevention of hypotension induced by spinal anesthesia in elective cesarean section. A systematic review and meta-analysis. Minerva Anestesiol. 2015 Sep;81(9):1019-30. Epub 2014 Dec 11. PMID 25501602
- [Result] Mercier FJ. Cesarean delivery fluid management. Curr Opin Anaesthesiol. 2012 Jun;25(3):286-91. doi: 10.1097/ACO.0b013e3283530dab. PMID 22459983
- [Result] Banerjee A, Stocche RM, Angle P, Halpern SH. Preload or coload for spinal anesthesia for elective Cesarean delivery: a meta-analysis. Can J Anaesth. 2010 Jan;57(1):24-31. doi: 10.1007/s12630-009-9206-7. Epub 2009 Oct 27. PMID 19859776
- [Result] Sharwood-Smith G, Drummond GB. Hypotension in obstetric spinal anaesthesia: a lesson from pre-eclampsia. Br J Anaesth. 2009 Mar;102(3):291-4. doi: 10.1093/bja/aep003. No abstract available. PMID 19218369
- [Result] Hwang J, Min S, Kim C, Gil N, Kim E, Huh J. Prophylactic glycopyrrolate reduces hypotensive responses in elderly patients during spinal anesthesia: a randomized controlled trial. Can J Anaesth. 2014 Jan;61(1):32-8. doi: 10.1007/s12630-013-0064-y. Epub 2013 Dec 18. PMID 24347351
- [Result] McDonnell NJ, Paech MJ, Muchatuta NA, Hillyard S, Nathan EA. A randomised double-blind trial of phenylephrine and metaraminol infusions for prevention of hypotension during spinal and combined spinal-epidural anaesthesia for elective caesarean section. Anaesthesia. 2017 May;72(5):609-617. doi: 10.1111/anae.13836. Epub 2017 Mar 3. PMID 28255987
- [Result] Cardoso MM, Yamaguchi ET, Amaro AR, Mezzetti R, Torres MA. Fetal and maternal effects of bolus of phenylephrine or metaraminol during spinal anesthesia for cesarean delivery. Anesthesiology. 2005;102:A31--A31.
- [Result] Abboud TK, Read J, Miller F, Chen T, Valle R, Henriksen EH. Use of glycopyrrolate in the parturient: effect on the maternal and fetal heart and uterine activity. Obstet Gynecol. 1981 Feb;57(2):224-7. PMID 7465128
- [Result] Ali-Melkkila T, Kaila T, Kanto J, Iisalo E. Pharmacokinetics of glycopyrronium in parturients. Anaesthesia. 1990 Aug;45(8):634-7. doi: 10.1111/j.1365-2044.1990.tb14385.x. PMID 2400072
- [Result] Mirakhur RK, Dundee JW. Glycopyrrolate: pharmacology and clinical use. Anaesthesia. 1983 Dec;38(12):1195-204. doi: 10.1111/j.1365-2044.1983.tb12525.x. PMID 6660460
- [Result] Ure D, James KS, McNeill M, Booth JV. Glycopyrrolate reduces nausea during spinal anaesthesia for caesarean section without affecting neonatal outcome. Br J Anaesth. 1999 Feb;82(2):277-9. doi: 10.1093/bja/82.2.277. PMID 10365009
- [Result] Quiney NF, Murphy PG. The effect of pretreatment with glycopyrrolate on emetic and hypotensive problems during caesarean section conducted under spinal anaesthesia. Int J Obstet Anesth. 2000;9:156-9.
- [Result] Chamchad D, Horrow JC, Nakhamchik L, Sauter J, Roberts N, Aronzon B, Gerson A, Medved M. Prophylactic glycopyrrolate prevents bradycardia after spinal anesthesia for Cesarean section: a randomized, double-blinded, placebo-controlled prospective trial with heart rate variability correlation. J Clin Anesth. 2011 Aug;23(5):361-6. doi: 10.1016/j.jclinane.2010.12.008. Epub 2011 May 31. PMID 21632228
- [Result] Yoon HJ, Cho HJ, Lee IH, Jee YS, Kim SM. Comparison of hemodynamic changes between phenylephrine and combined phenylephrine and glycopyrrolate groups after spinal anesthesia for cesarean delivery. Korean J Anesthesiol. 2012 Jan;62(1):35-9. doi: 10.4097/kjae.2012.62.1.35. Epub 2012 Jan 25. PMID 22323952
- [Result] Patel SD, Habib AS, Phillips S, Carvalho B, Sultan P. The Effect of Glycopyrrolate on the Incidence of Hypotension and Vasopressor Requirement During Spinal Anesthesia for Cesarean Delivery: A Meta-analysis. Anesth Analg. 2018 Feb;126(2):552-558. doi: 10.1213/ANE.0000000000002274. PMID 28704246
- [Result] Allen TK, George RB, White WD, Muir HA, Habib AS. A double-blind, placebo-controlled trial of four fixed rate infusion regimens of phenylephrine for hemodynamic support during spinal anesthesia for cesarean delivery. Anesth Analg. 2010 Nov;111(5):1221-9. doi: 10.1213/ANE.0b013e3181e1db21. Epub 2010 May 21. PMID 20495139
- [Result] Wang X, Mao M, Liu S, Xu S, Yang J. A Comparative Study of Bolus Norepinephrine, Phenylephrine, and Ephedrine for the Treatment of Maternal Hypotension in Parturients with Preeclampsia During Cesarean Delivery Under Spinal Anesthesia. Med Sci Monit. 2019 Feb 9;25:1093-1101. doi: 10.12659/MSM.914143. PMID 30738019
- [Result] Chabicovsky M, Winkler S, Soeberdt M, Kilic A, Masur C, Abels C. Pharmacology, toxicology and clinical safety of glycopyrrolate. Toxicol Appl Pharmacol. 2019 May 1;370:154-169. doi: 10.1016/j.taap.2019.03.016. Epub 2019 Mar 21. PMID 30905688
- [Result] Bruntion L (ed), Chabner B (ed), Knollman B (ed). Goodman & Gilman's The Pharmacological Basis of Therapeutics. 12th ed. New York: The McGraw Hill Companies; 2011.
- [Derived] Deshar R, Subedi A, Pokharel K, Sah BP, Prasad JN. Effect of glycopyrrolate on vasopressor requirements for non-elective cesarean section under spinal anesthesia: a randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2022 Oct 25;22(1):327. doi: 10.1186/s12871-022-01882-4. PMID 36284288